CLINICAL TRIAL: NCT00286221
Title: The Safety and Efficacy of IVPCA in the Management of Adult Postoperative Craniotomy Pain: A Prospective, Randomized Controlled Trial
Brief Title: IVPCA in the Management of Pain Following Major Intracranial Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00001283
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Intracranial Surgery
MeSH Terms: interventions — Passive Cutaneous Anaphylaxis; Fentanyl

STUDY DESIGN:
Who Masked: Care Provider

ARMS (4):
- Supratentorial PCA fentanyl (Experimental)
  Interventions: Drug: PCA fentanyl
- Supratentorial PRN fentanyl (Active Comparator)
  Interventions: Drug: PRN fentanyl
- Infratentorial PCA fentanyl (Experimental)
  Interventions: Drug: PCA fentanyl
- Infratentorial PRN fentanyl (Active Comparator)
  Interventions: Drug: PRN fentanyl

INTERVENTIONS:
Drug: PCA fentanyl — PCA fentanyl 0.5 ug/kg with a dosing interval ("lockout") of 15 minutes and a maximal permitted dosage of 4 demand doses per hour, according to their randomized preoperative assignment. The PCA pump (CADD-Solis Ambulatory Infusion Pump; Smiths Medical, Dublin, OH) had a preprogrammed dose limit of 50 ug fentanyl, and this was the maximal PCA dose permitted
  Other Names: PCA
  Arms: Infratentorial PCA fentanyl; Supratentorial PCA fentanyl
Drug: PRN fentanyl — IV fentanyl 25 to 50 ug every 30 minutes PRN (the maximal routine dose permitted in our Neurosciences Critical Care Unit (NCCU))
  Other Names: IV fentanyl
  Arms: Infratentorial PRN fentanyl; Supratentorial PRN fentanyl

SUMMARY:
This is a prospective, randomized controlled clinical trial to evaluate the efficacy and safety of intravenous patient controlled analgesia (IVPCA) in patients following major intracranial surgery (e.g. brain tumors, vascular surgery). We will compare pain, opioid consumption, costs, sedation level, length of hospital stay, patient satisfaction, and complications in patients randomized to receive either pro re nata (PRN) or IVPCA opioids. We hypothesize that IVPCA will be more efficacious than PRN opioids in the treatment of postoperative without an increased incidence of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing intracranial surgery

Exclusion Criteria:

* Patient refusal
* Pregnancy
* Aphasia
* Respiratory failure
* Allergy/intolerance to fentanyl
* Opioids use
* History of opioid-dependent pain,
* Patient has been in an investigational drug trial (except chemotherapy) in the month preceding the day of enrollment
* Mental or physical limitations that would prevent patient assessment or PCA use
* Chronic painful conditions unrelated to the reason for surgery,
* Clinically significant respiratory disease that required supplemental oxygen or ventilatory support such as use of mechanical ventilation or positive pressure ventilation
* Patient is unable to initiate a bolus dose of IVPCA fentanyl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradford Winters, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Result] Morad AH, Winters BD, Yaster M, Stevens RD, White ED, Thompson RE, Weingart JD, Gottschalk A. Efficacy of intravenous patient-controlled analgesia after supratentorial intracranial surgery: a prospective randomized controlled trial. Clinical article. J Neurosurg. 2009 Aug;111(2):343-50. doi: 10.3171/2008.11.JNS08797. PMID 19249923
- [Result] Morad A, Winters B, Stevens R, White E, Weingart J, Yaster M, Gottschalk A. The efficacy of intravenous patient-controlled analgesia after intracranial surgery of the posterior fossa: a prospective, randomized controlled trial. Anesth Analg. 2012 Feb;114(2):416-23. doi: 10.1213/ANE.0b013e31823f0c5a. Epub 2011 Dec 9. PMID 22156333

RESULTS

PARTICIPANT FLOW:
Groups:
- Supratentorial PCA Fentanyl: PCA fentanyl: Patient controlled analgesia (PCA) fentanyl 0.5 ug/kg with a dosing interval ("lockout") of 15 minutes and a maximal permitted dosage of 4 demand doses per hour, according to their randomized preoperative assignment. The PCA pump (CADD-Solis Ambulatory Infusion Pump; Smiths Medical, Dublin, OH) had a preprogrammed dose limit of 50 ug fentanyl, and this was the maximal PCA dose permitted
Period: Overall Study
Arm/Group | Supratentorial PCA Fentanyl | Supratentorial PRN Fentanyl | Infratentorial PCA Fentanyl | Infratentorial PRN Fentanyl
Started | 39 | 40 | 40 | 40
Completed | 29 | 35 | 31 | 34
Not Completed | 10 | 5 | 9 | 6
Not completed — Protocol Violation | 2 | 1 | 6 | 4
Not completed — Unanticipated Neurosurgical Complication | 6 | 3 | 3 | 2
Not completed — Inability to trigger PCA | 2 | 0 | 0 | 0
Not completed — Unrecognized exclusion criteria met | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Supratentorial PCA Fentanyl: PCA fentanyl: Patient controlled analgesia (PC fentanyl 0.5 ug/kg with a dosing interval ("lockout") of 15 minutes and a maximal permitted dosage of 4 demand doses per hour, according to their randomized preoperative assignment. The PCA pump (CADD-Solis Ambulatory Infusion Pump; Smiths Medical, Dublin, OH) had a preprogrammed dose limit of 50 ug fentanyl, and this was the maximal PCA dose permitted
- Supratentorial PRN Fentanyl: PRN fentanyl: IV fentanyl 25 to 50 ug every 30 minutes pro re nata (PRN) (the maximal routine dose permitted in our Neurosciences Critical Care Unit (NCCU))
- Total: Total of all reporting groups
Arm/Group | Supratentorial PCA Fentanyl | Supratentorial PRN Fentanyl | Infratentorial PCA Fentanyl | Infratentorial PRN Fentanyl | Total
Number analyzed (Participants) | 29 | 35 | 31 | 34 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (11.9) | 47.8 (15.0) | 45.4 (14.6) | 41.4 (11.1) | 45.6 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 20 | 21 | 76
  Male | 11 | 18 | 11 | 13 | 53
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 35 | 31 | 34 | 129

OUTCOME MEASURES:

1. Primary Outcome: Hourly Pain Scores
Description: Patients' Numerical Rating Scale scores (0-10: 0 = no pain, 10 = worst imaginable pain)
Time Frame: Up to 16 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supratentorial PCA Fentanyl | Supratentorial PRN Fentanyl | Infratentorial PCA Fentanyl | Infratentorial PRN Fentanyl
Number analyzed (Participants) | 29 | 35 | 31 | 34
units on a scale | 2.5 (2.0) | 3.6 (2.1) | 3.7 (1.9) | 5.2 (1.9)

2. Secondary Outcome: Fentanyl Consumption
Description: the amount of fentanyl is that administered in response to corresponding rest pain levels. Thus, the 0 hour indicates the amount of fentanyl administered from the time of admission until the end of the first hour. Also note that once pain assessments are made every other hour (e.g., 10, 12, 14, and 16), the analgesic totals indicated are for the corresponding 2-hour period after the pain assessment, and were halved to estimate the hourly rate of analgesic consumption.
Time Frame: Up to 16 hours
Measure: Mean (Standard Deviation); unit: mcg/hour
Arm/Group | Supratentorial PCA Fentanyl | Supratentorial PRN Fentanyl | Infratentorial PCA Fentanyl | Infratentorial PRN Fentanyl
Number analyzed (Participants) | 29 | 35 | 31 | 34
mcg/hour | 44.1 (34.5) | 23.6 (23.7) | 54.8 (34.8) | 29.9 (16.4)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected only during the time of patient enrollment in the study, up to 16 hours
Arm/Group | Supratentorial PCA Fentanyl | Supratentorial PRN Fentanyl | Infratentorial PCA Fentanyl | Infratentorial PRN Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/35 | 0/31 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/35 | 0/31 | 0/34
Other Adverse Events (participants affected / at risk) | 0/29 | 0/35 | 0/31 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes